CLINICAL TRIAL: NCT04505605
Title: Study of a Possible Respiratory Degradation Prognosis Caused by Biomarkers in Severe Forms of COVID-19 Pneumonia: the LPSARS2 Study
Brief Title: Study of a Possible Respiratory Degradation Prognosis Caused by Biomarkers in Severe Forms of COVID-19 Pneumonia
Acronym: LPSARS2
Status: Terminated | Type: Observational
Why Stopped: The PI decided to stop the study due to the low number of inclusions.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Centre Hospitalier Victor Dupouy (Other)
Responsible Party: Sponsor
Other Study IDs: LPSARS2
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Community-acquired Pneumonia; Covid19
Keywords: covid19; pneumonia; community acquired pneumonia; biomarkers
MeSH Terms: conditions — Community-Acquired Pneumonia; COVID-19; Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples on a dry tube with 5mL separating gel are collected, depending on patient hospitalization procedure.

GROUPS / COHORTS (3):
- Patient hospitalized without being transferred in the ICU: A blood sample on a dry tube with 5 ml separating gel in addition to the blood test made on the basis of the usual medical care, will be taken on D1 (day of the enrollment = the day of hospitalization in the healthcare institution). The total volume of blood collected as part of the research is therefore 5 ml.
  Interventions: Other: Blood samples
- Patient directly hospitalized in the ICU: A blood sample on a dry tube with a 5 ml separating gel in addition to the blood test made on the basis of the usual medical care, will be taken on D1 and D3 of the admission to intensive care. The total volume of blood collected for research is therefore 10 ml.
  Interventions: Other: Blood samples
- Patient transferred from an other hospital service to the ICU: A blood sample on a dry tube with 5 ml separating gel in addition to the blood test that will be taken at D1 and D3 of the patient's admission to the intensive care unit, even if it has already been included in the study during the patient's admission to the unit (D1 hospitalization). The total volume of blood collected for the research is therefore 15 ml.
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — A blood sample will be collected on a dry tube with 5mL separating gel on each enrolled patients. Those will be made depending on the patients hospitalization.

SUMMARY:
Respiratory infection with the SARS-CoV2 virus is associated with a major risk of viral pneumonia that can lead to respiratory distress requiring resuscitation. In the most severe forms, it may require a mechanical ventilation or even lead to an acute respiratory distress syndrome with a particularly poor prognosis. The SARS-CoV2 is a single-stranded RNA virus of positive polarity and belongs to the beta genus of Coronaviruses. SARS-CoV2 is responsible for the third epidemic in less than twenty years secondary to a Coronavirus (SARS-CoV then MERS-CoV) and if the mortality associated with it is lower than that of previous strains, particularly MERS-CoV (Middle East Respiratory Syndrome), its spread is considerably bigger. As a result, the number of patients developing respiratory distress that require an invasive mechanical ventilation is high, with prolonged ventilation duration in these situations.

DETAILED DESCRIPTION:
The mechanisms responsible for alveolar damage during viral pathologies, particularly Coronavirus, are very similar to those observed during acute respiratory distress syndromes in adults. Macrophages present in the pulmonary parenchyma appear to play a central role in the severity of the inflammatory response and the production of proinflammatory mediators, notably chemokines leading to secondary leukocyte infiltration. The recent monocytic origin could explain the particular severity of this inflammatory response whose usual control is no longer assured. The alteration of infectious control by alveolar macrophages during ageing also tends to confirm the central role of these cells in the pattern of respiratory distress observed during COVID-19 infection, which is particularly severe in the elderly.

In many situations, the endotoxin (or lipopolysaccharide, LPS) plays a major role in the pathophysiology and even the severity of respiratory damage, in particular, due to the existence of circulating endotoxin from the pathogenic agent responsible (Gram-negative bacteria), but also due to translocation of digestive origin in the context of sepsis (systemic inflammatory response) which is associated with (if not responsible for) respiratory aggression. Such an alteration of the mucous membrane is particularly noticeable in cases of obesity. The importance of this mechanism during pulmonary aggression of viral origin is, on the other hand, unknown.

Few data are available on the prediction of early onset of respiratory distress syndrome in low respiratory infection in the absence of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 18 years old
* French-speaking patient
* Patient whose COVID-19 respiratory infection was confirmed by laboratory tests (either by a PCR and any other commercial or public health tests) or a scanner, that requires a hospitalization in a healthcare institution.

Exclusion Criteria:

* Patient/ relative or proxy person opposed to the study participation
* Patient under guardianship or curators
* Patient deprived of liberty
* Patient under the safeguard of justice.
* Dying / Moribund patient
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged from 18 years, infected by the COVID-19 and suffers from a severe form of COVID 19 acquired pneumonia that requires an hospitalization.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of the dosage of biomarkers | 6 months = study duration
  The study aims at evaluating the interests of the biomarkers dosage: endotoxin (LPS) and circulating cytokines (HMGB1 or RAGE) in the prediction of respiratory degradation through a severe form of COVID-19 acquired pneumonia that requires a hospitalization.

SECONDARY OUTCOMES:
Link between the biomarkers | 6 months = study duration
  The study will be also focusing on the search for a correlation between the biomarkers by blood samples that will be taken on each hospitalized patients.

CONTACTS AND LOCATIONS:
Overall Officials: François PHILIPPART, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region